CLINICAL TRIAL: NCT02582398
Title: Influence of Light Exposure on Cerebral Monoamine Oxidase A in Seasonal Affective Disorder and Healthy Controls Measured by PET
Brief Title: Influence of Light Exposure on Cerebral MAO-A in Seasonal Affective Disorder and Healthy Controls Measured by PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Assoc. Prof. PD Dr. Rupert Lanzenberger, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 248/2011
Record Dates: First submitted 2015-06-04; First posted 2015-10-21 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Seasonal Affective Disorder
MeSH Terms: conditions — Seasonal Affective Disorder | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Light Therapy (Experimental): One subgroup of SAD patients and healthy controls respectively will receive bright light therapy using an artificial white light source (PhysioLight LD220 by DAVITA®, www.davita.de/shop/lichttherapiegeraete/lichtduschen-tageslicht/physiolight-ld-220.html) with full-spectrum 10.000lux light intensity. The treatment will be applied 30min per day at a distance of about of 50cm, preferably in the morning, during 3 weeks.
  Interventions: Other: Light Therapy
- Placebo Light (Placebo Comparator): The second subgroup of the SAD patients and healthy controls will receive a non-biologically active light source (<400nm or >500nm). Here, the lamp will have largely similar shape and size as compared to the therapeutic device, but the fluorescent tube with the high light intensity will be replaced by an ordinary bulb.
  Interventions: Other: Placebo Light

INTERVENTIONS:
Other: Light Therapy — One subgroup of SAD patients and healthy controls respectively will receive bright light therapy using an artificial white light source (PhysioLight LD220 by DAVITA®, www.davita.de/shop/lichttherapiegeraete/lichtduschen-tageslicht/physiolight-ld-220.html) with full-spectrum 10.000lux light intensity. The treatment will be applied 30min per day at a distance of about of 50cm, preferably in the morning, during 3 weeks.
  Arms: Light Therapy
Other: Placebo Light — The second subgroup of the SAD patients and healthy controls will receive a non-biologically active light source (<400nm or >500nm). Here, the lamp will have largely similar shape and size as compared to the therapeutic device, but the fluorescent tube with the high light intensity will be replaced by an ordinary bulb.
  Arms: Placebo Light

SUMMARY:
This study aims to assess differences in monoamine oxidase A (MAO-A) distribution in the brain between seasonal affective disorder patients and healthy controls using positron emission tomography. In addition the investigators aim to demonstrate the impact of light therapy on MAO-A distribution

In addition, a pilot study and a sub-study in healthy controls were performed

DETAILED DESCRIPTION:
This study aims to assess differences in monoamine oxidase A (MAO-A) distribution in the brain between seasonal affective disorder patients and healthy controls using positron emission tomography. In addition, the investigators aim to demonstrate the impact of light therapy on MAO-A distribution by investigating patients and controls in the winter before bright light therapy, in the winter after bright-light therapy, and in the summer. Bright light therapy will be placebo controlled, randomized, and double blinded.

ELIGIBILITY:
Inclusion Criteria for Patients:

* DSM-IV diagnosis of SAD established by diagnostic interview according to the SCID.
* Global Seasonality Score of 10 or higher on the Seasonal Pattern Assessment Questionnaire (SPAQ)
* Somatic health based on history, physical examination, ECG, and laboratory screening
* Aged 18 to 55 years
* No therapeutic treatment of SAD in the last 6 months (drugs and light therapy)
* Willingness and competence to complete the informed consent process

Inclusion criteria for healthy controls:

* Aged 18 to 55 years
* Somatic and psychiatric health based on history, physical examination, ECG, laboratory screening, SCID
* Willingness and competence to complete the informed consent process

Exclusion criteria for patients and healthy controls:

* Concomitant major medical or neurological illness
* Concomitant psychiatric disorders
* Current smoking
* Ingestion of antidepressants or other psychotropic agents targeting the serotonergic system, within the last 6 months.
* Bright light therapy within the last 6 months.
* Current substance abuse including alcohol, drugs of abuse, or any medication in a manner which is indicative of substance-related disorders (e.g. substance dependency) according to the DSM-IV.
* Failure to comply with the study protocol or follow the instructions of the investigators.
* Positive urine pregnancy test.
* For participants who participated in an earlier neuroimaging study using ionizing radiation, the total radiation exposure dose of 20 mSv over the last 10 years must not be exceeded, as specified in the legislation on radiation protection (Allg. Strahlenschutzverordnung 2010; www.ris.bka.gv.at).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2013-11; Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Change in MAO-A specific distribution volume (MAO-A DVs) assessed with PET | PET2 (3 weeks after PET1) compared to PET 1 (baseline), PET3 (6 months after PET1) compared to PET 1 (baseline) and PET 2 (3 weeks after PET1)

OTHER OUTCOMES:
Change in SAD symptoms assessed with Morningness-Eveningness-Questionnaire (MEQ) | PET2 (3 weeks after PET1) compared to PET 1 (baseline), PET3 (6 months after PET1) compared to PET 1 (baseline) and PET 2 (3 weeks after PET1)
Change in SAD symptoms assessed with Hamilton Depression Rating Scale with Atypical Depression Supplement (SIGH-ADS) | PET2 (3 weeks after PET1) compared to PET 1 (baseline), PET3 (6 months after PET1) compared to PET 1 (baseline) and PET 2 (3 weeks after PET1)
Change in SAD symptoms assessed with Beck Depression Inventory (BDI) | PET2 (3 weeks after PET1) compared to PET 1 (baseline), PET3 (6 months after PET1) compared to PET 1 (baseline) and PET 2 (3 weeks after PET1)
Light exposition assessed with photometer | During the 3 weeks of light therapy (between PET1 and PET2), 3 weeks before PET3
Difference in MAO-A specific distribution volume (MAO-A DVs) assessed with PET between patients and healthy controls | At PET1, PET2, and PET3

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Lanzenberger, MD, PD, A/Prof., Principal Investigator — Medical University of Vienna, Department of Psychiatry and Psychotherapy
Locations (1):
- Department of Psychiatry and Psychotherapy, Vienna, Austria

REFERENCES:
- [Derived] Schlosser G, Murgas M, Godbersen GM, Reichel S, Silberbauer L, Nics L, Winkler D, Stimpfl T, Hacker M, Kasper S, Rujescu D, Lanzenberger R, Spies M. Human in vivo assessment of ketamine binding of the serotonin transporter-follow up at a higher dose. Front Neurosci. 2025 Oct 2;19:1651016. doi: 10.3389/fnins.2025.1651016. eCollection 2025. PMID 41113438
- [Derived] Handschuh PA, Murgas M, Winkler D, Winkler-Pjrek E, Hartmann AM, Domschke K, Baldinger-Melich P, Rujescu D, Lanzenberger R, Spies M. Summer and SERT: Effect of daily sunshine hours on SLC6A4 promoter methylation in seasonal affective disorder. World J Biol Psychiatry. 2025 Apr;26(4):159-169. doi: 10.1080/15622975.2025.2477463. Epub 2025 Mar 20. PMID 40114401
- [Derived] Spies M, Murgas M, Vraka C, Philippe C, Gryglewski G, Nics L, Balber T, Baldinger-Melich P, Hartmann AM, Rujescu D, Hacker M, Winkler-Pjrek E, Winkler D, Lanzenberger R. Impact of genetic variants within serotonin turnover enzymes on human cerebral monoamine oxidase A in vivo. Transl Psychiatry. 2023 Jun 15;13(1):208. doi: 10.1038/s41398-023-02506-2. PMID 37322010
- [Derived] Handschuh PA, Murgas M, Vraka C, Nics L, Hartmann AM, Winkler-Pjrek E, Baldinger-Melich P, Wadsak W, Winkler D, Hacker M, Rujescu D, Domschke K, Lanzenberger R, Spies M. Effect of MAOA DNA Methylation on Human in Vivo Protein Expression Measured by [11C]harmine Positron Emission Tomography. Int J Neuropsychopharmacol. 2023 Feb 14;26(2):116-124. doi: 10.1093/ijnp/pyac085. PMID 36573644